CLINICAL TRIAL: NCT05660109
Title: A Double-blind, Randomized, Placebo-controlled, Phase 2a Study to Evaluate the Safety, Tolerability, and Pharmacodynamic (PD) Effects of Two Infusions of Escalating Doses of TPM502 in Adults Diagnosed With Celiac Disease
Brief Title: A Study to Assess the Safety of TPM502 in Adults With Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Topas Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCeD21
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Celiac Disease
Keywords: celiac disease; tolerance
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPM502 (Experimental)
  Interventions: Drug: TPM502
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TPM502 — TPM502 contains 3 peptides each consisting of two overlapping T cell epitopes that encompass the major gluten epitopes for HLA-DQ2.5
  Arms: TPM502
Other: Placebo — Placebo
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn about the safety and the pharmacodynamic (PD) effects of TPM502 in adults with celiac disease. The main questions it aims to answer are:

* if TPM502 is safe and well tolerated
* if TPM502 can induce modifications in parameters indicating that it may induce tolerance to gluten

Participants will:

* undergo 1-day gluten challenge during screening and after administration of TPM502 or placebo.
* receive 2 infusions of TPM502 or placebo, 2 weeks apart

DETAILED DESCRIPTION:
This is a multi center, double-blind, randomized, placebo-controlled Phase 2a study to evaluate the safety, tolerability, and PD effects of two infusions of TPM502 in adult patients diagnosed with CeD.

The patient´s participation in the study comprises 3 phases: screening period, treatment period and follow-up period.

Patients fulfilling the eligibility criteria will be randomized to receive two infusions of TMP502 (or placebo) at the same dose level. Patients will undergo a second GC one week after the second infusion of TPM502.

The study includes 4 cohorts of patients, each cohort will receive escalating doses of TPM502 (or placebo). Upon completion of the 3rd cohort, a lower dose can be investigated, if deemed relevant.

ELIGIBILITY:
Inclusion Criteria:

* Availability of a documented biopsy-confirmed diagnosis of CeD OR documented tissue transglutaminase >10x ULN and documented positive IgA anti-endomysial antibody (EMA) at time of CeD diagnosis (as per local guidelines)
* Serum anti-tissue transglutaminase 2 immunoglobin A antibodies within normal range (i.e., <15 U/mL) at screening
* Serum IL-2 levels (AUC1-6h) above a pre-defined threshold following the GC at screening
* Patients must have been on GFD for ≥ 6 months
* Patients must have well-controlled CeD, defined as mild or with no ongoing signs or symptoms felt to be related to active CeD, as per investigator's assessment
* HLA-DQ2.5 positive

Exclusion Criteria:

* Known or suspected refractory CeD (refractory CeD type I or II)
* Known intolerable symptoms following previous GCs, as per investigator's assessment
* HLA DQ8 positive
* Any active gastrointestinal disease such as gastroesophageal reflux disease, esophagitis or peptic ulcer, microscopic colitis, or irritable bowel syndrome, which in the opinion of the investigator might interfere with the assessment of the symptoms related to CeD
* Known history of or active Crohn's disease, ulcerative colitis, or ulcerative jejunitis
* Known wheat allergy
* Known hypersensitivity to i.v. iron preparations or any other excipients present in the reconstituted TPM502 or placebo

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, causality, and outcomes of treatment-emergent adverse events | throughout the study, on average 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Knut Lundin, MD, Principal Investigator — Oslo University Hospital
Locations (8):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide
  - Wesley Research Institute, Brisbane
- CRST Oy, Turku, Finland
- Charite' Hospital, Berlin, Germany
- Centre for Human Drug Research, Leiden, Netherlands
- Norway (2):
  - Oslo University Hospital HF - Rikshospitalet, Oslo
  - University Hospital of North-Norway, Tromsø
- Clinical Trial Consultants, Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No